CLINICAL TRIAL: NCT05685472
Title: A Phase 1, Open-label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Antitumor Activity of MEDI5752 in Japanese Subjects With Advanced Solid Tumors
Brief Title: MEDI5752 in Japanese Patients With Advanced Solid Tumors.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D7980C00006
Record Dates: First submitted 2022-11-09; First posted 2023-01-17 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced Solid Tumors; Phase1; Safety; Tolerability; Pharmacokinetics; Immunogenicity; Antitumor Activity; MEDI5752

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MEDI5752 monotherapy (Experimental)
  Interventions: Biological: MEDI5752

INTERVENTIONS:
Biological: MEDI5752 — Subjects will remain on treatment until unacceptable toxicity, documentation of progressive disease, or development of other reason for treatment discontinuation.

SUMMARY:
This is a Phase 1, open-label study evaluate the safety, tolerability, pharmacokinetics, immunogenicity and anti-tumor activity of MEDI5752 in Japanese patients with advanced solid solid tumors.

DETAILED DESCRIPTION:
<Objectives>

Primary Objective:

To evaluate the safety and tolerability of MEDI5752 in Japanese subjects with advanced solid tumors.

Secondary Objective:

To assess the anti-tumor activity and efficacy of MEDI5752. To describe the pharmacokinetics of MEDI5752.

Exploratory Objective:

To conduct exploratory research into factors that may be predictive of response or may influence the progression of cancer and/or response (efficacy) to MEDI5752.

Eligible patients will be administered as a single dose at each Cycle Day1. Each cycle from Cycle 1 has a duration of 21 days.

A minimum of 3 and a maximum of 9 evaluable patients will be enrolled in each cohort.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 18 years at the time of screening
2. World Health Organization/Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at enrollment
3. Life expectancy ≥ 12 weeks
4. Histologically or cytologically-confirmed advanced solid tumors
5. Subjects who have received prior anti-PD-1, anti-PD-L1, or anti-CTLA-4 therapy or any concurrent chemotherapy, radiotherapy, investigational, biologic, or hormonal therapy for cancer treatment may be eligible to enter the study following a washout period as applicable
6. Females of childbearing potential who are sexually active with a nonsterilized male partner must use at least one highly effective method of contraception
7. Nonsterilized males who are sexually active with a female partner of childbearing potential must use a male condom from Day 1 and for 90 days after the final dose of investigational product.
8. Subjects must have at least one measurable lesion
9. Adequate organ and marrow function
10. Signed and dated written informed consent
11. Subjects must provide tumor material as applicable

Exclusion Criteria

1. Involvement in the planning and/or conduct of the study (applies to both sponsor staff and/or staff at the study site)
2. Concurrent enrollment in another clinical study, unless it is an observational clinical study or the follow-up period of an interventional study
3. For subjects who have received prior anti-PD-1, anti-PD-L1, or anti-CTLA-4:

   1. Subjects must not have received anti-PD-1, anti-PD-L1, anti-CTLA-4 or any other immunotherapy or immune-oncology (IO) agent within 21 days of commencing treatment with investigational product.
   2. Subject must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy.
   3. All AEs while receiving prior immunotherapy must have completely resolved or resolved to Grade 1 prior to screening for this study.
4. Current or prior use of immunosuppressive medication within 14 days before the first dose of investigational product is excluded.
5. Receipt of live attenuated vaccine within 30 days prior to the first dose of investigational product.
6. Active or prior documented autoimmune or inflammatory disorders
7. History of organ transplant
8. Known allergy or reaction to any component of the planned study treatment.
9. Untreated CNS metastatic disease, leptomeningeal disease, or cord compression
10. Unresolved toxicities from prior anticancer therapy, defined as having not resolved to NCI CTCAE v5.0 Grade 0 or 1, or to levels dictated in the inclusion/exclusion criteria
11. Major surgical procedure (as defined by the investigator) within 28 days prior to the first dose of Investigational Product or still recovering from prior surgery
12. Female subjects who are pregnant or breastfeeding, as well as male or female subjects of reproductive potential who are not willing to employ one highly effective method of birth control
13. Uncontrolled intercurrent illness, that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the subject to give written informed consent.
14. Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of the subject's safety or study results
15. Judgment by the investigator that the subject is unsuitable to participate in the study and the subject is unlikely to comply with study procedures, restrictions, and requirements.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-12-08 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
The number of subjects experiencing treatment related adverse events (AEs) | From the time of informed consent through 90 days following termination of treatment with investigational product
  The primary endpoint is as assessed by the number of subjects experiencing adverse events (AEs) graded per NCI CTCAE v5.0.
The number of subjects experiencing treatment related serious adverse events (SAEs) | From the time of informed consent through 90 days following termination of treatment with investigational product
  The primary endpoint is as assessed by the number of subjects with serious adverse events (SAEs) graded per NCI CTCAE v5.0.
The number of subjects experiencing dose-limiting toxicities (DLTs) | Up to 21 days following the first dose
  The primary endpoint is as assessed by the number of subjects experiencing dose limiting toxicities (DLTs) as defined by the protocol.
The number of subjects experiencing abnormal laboratory evaluations | From the time of informed consent through 90 days following termination of treatment with investigational product
  The primary endpoint is as assessed as the number of subjects experiencing changes in laboratory parameters from baseline.
The number of subjects experiencing changes from baseline in vital signs reported as adverse events | From the time of informed consent through 90 days following termination of treatment with investigational product
  The primary endpoint is as assessed by the number of subjects experiencing clinically significant changes in vital signs from baseline.
The number of subjects experiencing abnormal electrocardiograms (ECG) reported as Adverse Events | From the time of informed consent through 90 days following termination of treatment with investigational product
  The primary endpoint is as assessed by the the number of subjects experiencing clinically significant changes in ECG parameters from baseline.

SECONDARY OUTCOMES:
Preliminary anti-tumor activitiy of MEDI5752 using Objective Response based on RECIST v1.1 | From the first dose of study drug through the date of documented progression, end of study, or date of death until study completion assessed up to 16 months.
  The endpoints for assessment of antitumor activity is defined by using ORR, PFS, BOR,DCR, DoR and TTR according to RECIST v1.1.
Pharmacokinetics of MEDI5752 | At Cycle1Day1, ,Cycle1Day2, Cycle1Day3, Cycle1Day8, Cycle1Day15, Cycle2Day1, Cycle2Day8, Cycle3Day1, Cycle4Day1, Cycle5Day1, Cycle6Day1, Cycl7Day1, every 6 weeks after Cycle7Day1 (each cycle is 21 days) and up to 90 days following end of treatment.
  The endpoints for the assessment of PK of MEDI5752 include individual MEDI5752 concentrations at different time points after administration. (e.g., Maximum plasma concentration[Cmax]）
Immunogenicity of MEDI5752 | At Cycle1Day1, Cycle1Day8, Cycle1Day15, Cycle2Day1, Cycle2Day8, Cycle3Day1, Cycle4Day1, Cycle5Day1, Cycle6Day1, Cycl7Day1, every 6 weeks after Cycle7Day1 (each cycle is 21 days) and up to 90 days following end of treatment.
  The endpoints for the immunogenicity of MEDI5752 include the number of subjects who develop detectable anti-drug antibodies (ADAs)
PD-L1 Expression in subjects with advanced solid tumors | To be assessed at at baseline
  The endpoint for the PD-L1 expression will be determined by Immunohistochemistry characterization.

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Research Site, Chūōku
  - Research Site, Kashiwa

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home